CLINICAL TRIAL: NCT05922930
Title: Phase I/II Study of TROP2 CAR Engineered IL15-transduced Cord Blood-derived NK Cells Delivered Intraperitoneally for the Management of Platinum Resistant Ovarian Cancer, Mesonephric-like Adenocarcinoma, and Pancreatic Cancer
Brief Title: Study of TROP2 CAR Engineered IL15-transduced Cord Blood-derived NK Cells Delivered Intraperitoneally for the Management of Platinum Resistant Ovarian Cancer, Mesonephric-like Adenocarcinoma, and Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0687; NCI-2023-05027 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer; Ovarian Cancer; Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Ovarian Neoplasms; Adenocarcinoma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TROP2-CAR-NK (Experimental): Participants will receive 1 dose of TROP2-CAR-NK and will visit the study clinic up to 16 times to have tests and procedures (such as blood draws, biopsies, and CT scans).
  Participants will receive lymphodepleting chemotherapy (cyclophosphamide and fludarabine) for 3 days in a row. Participants will receive cyclophosphamide and fludarabine by vein over about 3 hours total.
  Interventions: Drug: TROP2-CAR-NK; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: TROP2-CAR-NK — Given by IP (intraperitoneal)
Drug: Cyclophosphamide — Given by IV (vein)
Drug: Fludarabine — Given by IV (vein)

SUMMARY:
To find the recommended dose of TROP2- CAR-NK given intraperitoneally (directly into the abdominal cavity) to patients with highgrade serous ovarian cancer that has not responded to previous treatment or is resistant to treatment.

DETAILED DESCRIPTION:
Primary Objectives:

1. To determine the safety and optimal cell dose of TROP2-CAR/IL15-transduced CB-NK cells[TROP2-CAR NK cells (KSR)]delivered intraperitoneally and define the MTD/RP2D.

Endpoints

1. Dose-limiting toxicity
2. MTD and RP2D of TROP2-CAR/IL15-transduced CB-NK cells and TROP2-CAR/IL15-transduced CB-NK cells [TROP2-CAR NK cells (KSR)] dose

Secondary Objectives and Endpoints

Objectives:

1. To estimate the best objective response rate (ORR) in patients at 12 weeks after infusion.
2. To estimate median progression free survival.
3. To quantify persistence of infused allogeneic donor CAR-transduced CB-derived NK cells in the peripheral blood and peritoneal cavity in the recipient.
4. To profile and assess the dynamic changes in the peritoneal tumor microenvironment before and after treatment using single-cell transcriptional and immune profiling on peritoneal cells at various time points before and after treatment.
5. To estimate patient reported symptom burden and quality of life longitudinally through treatment and follow up.
6. To compare changes in circulating tumor DNA (ctDNA) with response as determined by RECIST v1.1

Endpoints:

1. Objective response rates at week 12
2. Median progression free survival
3. TROP2-CAR NK cell numbers in peripheral blood and peritoneal cavity vs time profile
4. Characterization of lymphocyte populations at various time points
5. PROMIS-19, EQ-5D-5L, and MDASI-OC PRO questionnaire responses
6. Plasma ctDNA concentration at baselines and serial timepoint

ELIGIBILITY:
Inclusion criteria:

1. Subjects must be 18 years or older.
2. Subjects must be willing and able to provide informed consent.
3. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. A female participant is eligible to participate if at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 1
   2. A WOCBP who agrees to follow the contraceptive guidelines in Appendix 1 during the treatment period and for at least 3 months after the last dose of study treatment.
5. Subjects must have measurable disease present as defined by modified RECIST v1.1 criterion, and have disease present in the peritoneal cavity or retroperitoneal lymph nodes. Disease outside the peritoneal cavity is allowed as long as metastases are present within the peritoneal cavity or retroperitoneum.
6. Subject tumors must demonstrate at least 1+ TROP2 expression by immunohistochemistry.
7. Subjects must be at least 3 weeks from last cytotoxic chemotherapy at the time of starting lymphodepleting chemotherapy.
8. Subjects must be willing to undergo intraperitoneal port placement and scheduled peritoneal fluid and peripheral blood draws.
9. Subjects must have adequate organ function as defined in the following table (Table 1). Specimens must be collected within 10 days prior to the start of study treatment.

Table 1. Adequate Organ Function Laboratory Values Systemic Function Test Laboratory Value Hematologic Absolute neutrophil count (ANC) ≥1500/µL Platelets ≥100,000/µL Hemoglobin ≥8.0 g/dL (transfusion is allowed)a Renal Creatinine OR Creatinine clearance (CrCl) by Cockroft-Gault

* 1.5 x ULNb

  * 30 mL/min for participants with creatinine > 1.5 x ULNb Hepatic Total bilirubin ≤1.5 x ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 x ULN AST (SGOT) and ALT (SGPT) ≤2.5 x ULN (≤5 x ULN for participants with liver metastases) Coagulation International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 x ULN unless participate is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants ALT (SGPT) = alanine aminotransferase (serum glutamic pyruvic transaminase);AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.

    1. Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks of the screening test. Participants may be on a stable dose of erythropoietin (≥ approximately 3 months).
    2. Serum creatinine and creatinine clearance (CrCl) should be interpreted and calculated per institutional standard.

       Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.

       Inclusion Criteria:

       Ovarian Cancer:
       1. Subjects must have a histology confirming diagnosis of high grade serous ovarian/peritoneal/fallopian tube cancer with pathology reviewed at MD Anderson Cancer Center.
       2. Subjects must have failed at least two prior lines of chemotherapy (i.e. frontline adjuvant chemotherapy plus one additional line for recurrent/progressive disease), or have platinumresistant disease defined as disease progression on a platinum-containing agent or recurrence within 180 days of prior dose of a platinum-containing chemotherapeutic regimen.
       3. To be eligible, germline/somatic BRCA1/2 mutation carriers should have received prior PARPi therapy.

          Mesonephric-like adenocarcinoma:

       <!-- -->

       1. A histology confirming diagnosis of mesonephric-like adenocarcinoma (MLA) originating from the female reproductive tract or peritoneal lining (including MLA arising from endometriosis) with pathology reviewed at MD Anderson Cancer Center.
       2. Subjects must have failed at least one prior line of platinum-containing chemotherapy.

          Pancreatic Cancer:

       <!-- -->

       1. Subjects with histologically confirmed diagnosis of pancreatic ductal adenocarcinoma or ampullary-type carcinoma
       2. Subjects who have progressive disease after receiving initial treatment with either FOLFIRINOX, and/or a gemcitabine-based therapy

          Exclusion Criteria:

       <!-- -->

       1. Pregnant, breastfeeding, or expecting to conceive within the projected duration of the study, starting with the screening visit through 3 months after the last dose of trial treatment.

          If a WOCBP has a positive urine pregnancy test within 72 hours prior to hospital admission that cannot be confirmed as negative, a serum pregnancy test will be required (see Appendix 1).
       2. Has received systemic anti-cancer therapy including investigational agents within 4 weeks of starting lymphodepleting chemotherapy.
       3. Participants must have recovered from all AEs due to previous therapies to ≤ Grade 1 or baseline.

          Participants with ≤ Grade 2 neuropathy, alopecia, or other non-relevant AEs may be deemed eligible at the discretion of the PI. If a participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
       4. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
       5. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine.

          Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; However, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
       6. Is currently receiving another investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention. Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
       7. Diagnosis of immunodeficiency or receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
       8. History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in-situ cancers.
       9. Known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
       10. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is allowed.
       11. History of interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
       12. Active infection requiring systemic therapy.
       13. Known history of uncontrolled Human Immunodeficiency Virus (HIV) infection. Patients with HIV infection and undetectable viral load may participate.
       14. Known history of chronic Hepatitis B or Hepatitis C virus infection.
       15. Known history of active TB (Bacillus Tuberculosis).
       16. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
       17. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
       18. Has had an allogenic tissue/solid organ transplant.
       19. Clinically significant cardiovascular disease within 12 months from first dose of study intervention, including New York Heart Association (NYHA) Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular event, or cardiac arrhythmia associated with hemodynamic instability. Note: medically controlled arrhythmia would be permitted.
       20. Prolongation of QTcF interval to >480 ms
       21. Bleeding or thrombotic disorders or subjects at risk for severe hemorrhage. Subject with known deep vein thrombosis/pulmonary embolism that are under appropriate anti-coagulation treatment are eligible.
       22. Radiographic evidence of tumor encasement or invasion of a major blood vessel, or intra-tumoral cavitation.
       23. Active peritonitis or diverticulitis
       24. Medical or surgical history that in the treating physician's opinion would make the subjective not a suitable candidate for intraperitoneal therapy. Examples would include surgically documented extensive intraperitoneal adhesions or large volume ascites.
       25. History of severe hypersensitivity reaction with biologic therapy (e.g. monoclonal antibodies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amir Jazaeri, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org